CLINICAL TRIAL: NCT05382260
Title: Can Personal Music Change the Functional Connectivity of Disorders of Consciousness
Brief Title: Personal Music for Disorders of Consciousness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qiuyou Xie (Other)
Responsible Party: Sponsor-Investigator, Qiuyou Xie, principal investigator, Zhujiang Hospital
Organization: Zhujiang Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L20220318
Record Dates: First submitted 2022-04-01; First posted 2022-05-19 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Disorder of Consciousness
Keywords: DOC; preferred music; functional connectivity
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disorders of consciousness(DOC) (Experimental): The participants in this arm are disorders of consciousness, containing of vegetative state(VS) and minimally conscious state(MCS).
  Interventions: Other: Listening to music
- Health control (Other): They are health people with normal hearing, acting as a control for DOC group.
  Interventions: Other: Listening to music

INTERVENTIONS:
Other: Listening to music — After 5 minutes baseline, participants would listen to three kinds of music with 3 minutes washout and another 5 minutes baseline in the end, while EEG would record their cortical activity. And the order of the three kinds of music is random.

SUMMARY:
Background: The evaluation and treatment of disorders of consciousness(DOC) is a challenging undertaking. Now many neuroimaging techniques were used to detect the level of consciousness and electroencephagram(EEG) was widely used because of its high temporal resolution. Music would be an effective for DOC, due to its highly arousal value. Preferred music was near to persons, so that it would excite more range of cortical and increase the functional connectivity between cortices.

Methods: The exploratory study included 15 health controls and 30 DOC, with 15 minimally conscious state(MCS) and 15 vegetative state(VS). After 5 minutes baseline silence, they listened to relaxing music(RM), preferred music(PM) and amplitude modulated sound(AMS), with 5 minutes baseline silence in the end, meanwhile EEG recorded their cortical activity. Each music was appropriately 5 minutes and separated by 3 minutes washout.

Discussion: The study would verify the effect of preferred music to the functional connectivity of DOC. Music would excite the networks related to consciousness by cross-modal.

ELIGIBILITY:
Inclusion Criteria:

1. being DOC less than 1 year and more than 28 days;
2. diagnosis of VS and MCS based on CRS-R;
3. the auditory sub-scale of CRS-R scoring more than 0, or Auditory Brainstem Response showing no auditory injury at least one side;
4. stopping using sedatives more than 24 hours prior to study;
5. no history of neurological or psychiatric diseases.

Exclusion Criteria:

1. Auditory Brainstem Response showing completely injured auditory pathway(disappeared wave Ⅴ);
2. having epilepsy or EEG showing alpha-coma;
3. widely range of injured scalp or bone.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional connectivity for Baseline EEG | After approximately 5 minutes baseline.
  EEG would record participants' cortical activity while they are keeping quiet with their eyes opened for 5 minutes, and parameters relative to functional connectivity which could be calculated from offline EEG data. The EEG data would be separated to five frequency bands: δ (1-4 Hz), θ (4-8 Hz), α (8-13 Hz), β (13-30 Hz), and γ (30-45 Hz) and the functional connectivity would be calculated by each frequency bands.
Functional connectivity for relaxing music EEG | After approximately 5 minutes relaxing music.
  EEG would record participants' cortical activity while they are listening to relaxing music for approximately 5 minutes, and parameters relative to functional connectivity which could be calculated from offline EEG data. The EEG data would be separated to five frequency bands: δ (1-4 Hz), θ (4-8 Hz), α (8-13 Hz), β (13-30 Hz), and γ (30-45 Hz) and the functional connectivity would be calculated by each frequency bands.
Functional connectivity for preferred music EEG | After approximately 5 minutes preferred music.
  EEG would record participants' cortical activity while they are listening to preferred music for approximately 5 minutes, and parameters relative to functional connectivity which could be calculated from offline EEG data. The EEG data would be separated to five frequency bands: δ (1-4 Hz), θ (4-8 Hz), α (8-13 Hz), β (13-30 Hz), and γ (30-45 Hz) and the functional connectivity would be calculated by each frequency bands.
Functional connectivity for amplitude modulated sound EEG | After approximately 6 minutes amplitude modulated sound.
  EEG would record participants' cortical activity while they are listening to amplitude modulation sound for approximately 6 minutes, and parameters relative to functional connectivity which could be calculated from offline EEG data. The EEG data would be separated to five frequency bands: δ (1-4 Hz), θ (4-8 Hz), α (8-13 Hz), β (13-30 Hz), and γ (30-45 Hz) and the functional connectivity would be calculated by each frequency bands.

SECONDARY OUTCOMES:
Heart Rate Variability(HRV) for baseline | After approximately 5 minutes baseline.
  Another two electrodes would be placed upon the hands and record participants' heart rate. HRV would be analyzed offline.
Heart Rate Variability(HRV) for relaxing music | After approximately 5 minutes relaxing music.
  Another two electrodes would be placed upon the hands and record participants' heart rate. HRV would be analyzed offline.
Heart Rate Variability(HRV) for preferred music | After approximately 5 minutes preferred music.
  Another two electrodes would be placed upon the hands and record participants' heart rate. HRV would be analyzed offline.
Heart Rate Variability(HRV) for amplitude modulated sound | After approximately 6 minutes amplitude modulated sound.
  Another two electrodes would be placed upon the hands and record participants' heart rate. HRV would be analyzed offline.
The Music Therapy Assessment Tool for Awareness in Disorders of Consciousness(MATADOC) | After approximately 5 minutes preferred music.
  A scale contains three sub-scale, such as Principal Subscale: Essential Categories(scoring from 0 to 17, with the higher scores, the better status), Musical parameter and behavioural response type(scoring from 13 to 26, with the higher scores, the better status), Clinical information to inform goal setting and clinical care. The music therapist would give score from watching the video after study.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China